CLINICAL TRIAL: NCT05766072
Title: 5 Year- Follow up of Anxious and Sad Children
Brief Title: Early Intervention Coping Kids (TIM) Follow up Study
Acronym: FOPPT4
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: The Dam Foundation (Other)
Responsible Party: Principal Investigator, Kristin Martinsen, Principal Investigator, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 426598
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Anxiety Disorders; Depression
Keywords: Anxiety; Depression; School absenteeism; Youth
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Active Comparator): Youth in this arm received the intervention over 10 weeks during one semester (recruiting children over 6 semesters in total), children meeting in groups of approx. seven children. The groups were led by school health nurses.
  At the same time parents met for 7 group sessions, with the children participating in four of these
  Interventions: Other: EMOTION Kids coping with anxiety and depression (Mestrende barn in Norwegian)
- Control arm (No Intervention): The youth in the control condition received treatment as usual, e.g. talks with school health nurses or no intervention

INTERVENTIONS:
Other: EMOTION Kids coping with anxiety and depression (Mestrende barn in Norwegian) — The intervention is transdiagnostic and based on cognitive behavioral therapy where the children and their parents meet i groups led of school health nurses. They are learning coping skills to meet challenging and avoided situations, learning about emotion regulation, physical symptoms conitive restructuring and exposure/behavioral activation. Te manual is publshed in a US/English version and in a Norwegian version.
  Arms: Intervention arm

SUMMARY:
The project objectives are to investigate if a preventive intervention targeting anxious and sad children aged 8 to 12 years has haf the anticipated long-term effects, 5 years after receiving the intervention. Hence: will an indicated intervention reduce the incidence of common mental disorders in youth in the long term? The current study is a 5 year follow up of the previously completed RCT called the TIM-study (Clinical Trials identifier: NCT 02340637).

The aim of this study is to determine the long-term effects of the intervention to examine if true preventive effects are achieved as indicated by lower symptom levels, better functioning og fewer diagnosis of anxiety and depression 5 years after receiving an indicated preventiv intervention.

ELIGIBILITY:
Inclusion Criteria:

* Participants who participated in the previous randomized controlled TIM study (children then aged 8- 12 years selfreporing elevated symptom levels of anxiety and/or depression)

Exclusion Criteria:

* all earlier participats from the TIM study may enter the follow up study
* participants who chose to not participate in the 5-year follow-up of the TIM study are excluded from the follow-up study.

Ages: 13 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 450 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Multidimensional anxiety scale for children | 5- year follow up
  This 39-item, child self-report, assesses anxiety in youth ages 8 - 19, 0 - 117, higher score, higher anxiety
The Mood and Feelings Questionnaire Short version | 5-year follow up
  SMFQ comprised of 13 questions assessing cognitive, affective and behavioral-related depressive symptoms in youth ages 8 - 18 during the last two weeks, 0 - 26, higher score indicating higher levels of depression
The ADIS (Anxiety Disorders Interview Schedule) | 5-year follow up
  Relevant sections of this semi-structured interview (anxiety and depression), categorical outcome, have diagnosis/does not have diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Jo Magne Ingul, PhD, Principal Investigator — Regional Centre for Child and Youth Mental Health and Child Welfare (RKBU), Trondheim, Norway; Frode Adolfsen, PhD, Principal Investigator — Regional Centre for Child and Youth Mental Health and Child Welfare North, UiT, Tromsø, Norway
Locations (1):
- University of Oslo, Oslo, Norge, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Angold, A., Costello, E. J., Messer, S. C., & Pickles, A. (1995). Development of a short questionnaire for use in epidemiological studies of depression in children and adolescents. International Journal of Methods in Psychiatric Research, 5(4), 237-249.
- [Background] Kendall, P. C., Stark, K. D., Martinsen, K., O'Neil, K. A., & Arora, P. (2013). EMOTION:
- [Background] March, J. S. (1997). MASC - Multidimensional Anxiety Scale for Children - Technical Manual. Toronto, Canada: Multi-Health Systems.
- [Background] Martinsen, K. D., Kendall, P. C., Stark, K. D., Rodriguez, K. A. O. N., & Arora, P. (2014). Mestrende barn, gruppeledermanual barn. Oslo, Norway: Gyldendal Akademisk.
- [Background] Patras J, Martinsen KD, Holen S, Sund AM, Adolfsen F, Rasmussen LP, Neumer SP. Study protocol of an RCT of EMOTION: An indicated intervention for children with symptoms of anxiety and depression. BMC Psychol. 2016 Sep 26;4(1):48. doi: 10.1186/s40359-016-0155-y. PMID 27671742
- [Background] Silverman, W. K., Albano, A.M. Anxiety Disorders Interview Schedule (ADIS-IV): Child Interview Schedules. Oxford University Press, 2010).